CLINICAL TRIAL: NCT04565782
Title: Corona Virus Infection Among Liver Transplant Recipients: A Multicenter Study
Brief Title: Corona Virus Infection Among Liver Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dr. Nahed A. Makhlouf, Professor of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: 17300475
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: SARS-CoV Infection; Corona Virus Infection; Liver Transplant Recipient; COVID-19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A new strain of coronavirus that caused severe respiratory disease in infected individuals was initially identified in China's Wuhan City in December 2019. Severe acute respiratory distress syndrome coronavirus-2 (SARS-CoV-2), which was responsible for the corona virus infectious disease-2019 (COVID-19).The World Health Organization declared that COVID-19 was a Public Health Emergency of International Concern on January 30,2020.

The impact of COVID-19 in liver recipients remains largely unknown but accumulating experience is going on.

Liver transplant recipients should have been classified as a risk group and should have received regular surveillance for COVID-19 throughout the pandemic.

Some reports suggest decreasing immunosuppression for infected recipients, if no recent rejection episodes. Paradoxically, others suggest that a reactive immune response might be the cause for severe tissue damage, and that immunosuppression might be protective from the postulated cytokine storm.

Some studies stated that the LT patients who are permanently on immunosuppressants could be particularly susceptible to SARS-CoV-2, and their prognosis could be worse in comparison to the normal population. They recommended that LT recipients should be closely monitored for SARS-CoV-2.

The LT society of India (LTSI) highlighted the potential of LT recipients as asymptomatic carriers and source of viral spread, and that SARS-CoV-2 can be transmitted to LT recipients. There are insufficient data on the relationship between immunosuppressive therapy and COVID-19 in LT recipients during this pandemic. However, the Beijing working party for liver transplantation suggested that LT recipients who were infected with SARS-CoV-2 should be treated with steroids for a short period to reduce the severity of pneumonia.

They also suggested that immunosuppressive therapies should be continued for both patients with mild COVID-19 and those who were not infected by the virus, and calcineurin inhibitor treatment dosage should be reduced in moderate to severe cases.

Neutralizing antibodies (NAbs) play an important role in virus clearance and have been considered as a key immune product for protection or treatment against viral diseases. Virus-specific NAbs, induced through either infection or vaccination, have the ability to block viral infection. SARS-CoV -2 specific NAbs reached their peak in patients from day 10-15 after the onset of the disease and remained stable thereafter in the patients. Antibodies targeting on different domains of S protein, including S1, RBD, and S2, may all contribute to the neutralization.

Al-Rajhi Liver Center is the only liver transplantation center in Upper Egypt that performed only 51 living donor liver transplantation (LDLT) cases since 2014, but it was used as isolation Hospital for COVID-19 cases from March to July, 2020. Communication with liver transplant cases during that period was via Telemedicine. Resuming usual Hospital activity as Tertiary Liver Center occurred in 15 August 2020. Similarly, other Hospitals in Egypt were designated as COVID-19 isolation Hospitals.

DETAILED DESCRIPTION:
1. Liver Transplant recipients in 3 liver transplant centers will answer survey including 21 questions (14 questions covers the demographic data, date since the operation and immunosuppressant medications and 11 questions related to Corona virus infection). (SARS-CoV-2 infection will be defined according to the Ministry of Health and population definitions of suspected and confirmed cases).
2. Doing serological test searching for Neutralizing Ab against SARS-Corona virus 2 in the liver transplant recipients who accepted to give blood sample.

(It can be detected by Electrochemiluminescence immunoassay (ECLIA) method.

ELIGIBILITY:
Inclusion Criteria:

-Liver transplant recipients in 3 Liver Transplant Centers in Egypt and who accept to participate in the study

Exclusion Criteria:

* Those who refuse to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Liver transplant recipients in 3 Liver Transplant Centers in Egypt and who accept to participate in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of corona virus infection (confirmed or suspected) among liver transplant recipients | 1 month

SECONDARY OUTCOMES:
The presence of Neutralizing Ab against SARS-Corona virus 2 among liver transplant recipients whether who give symptoms for corona virus or asymptomatic and who accept to give blood sample | 2 month

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt